CLINICAL TRIAL: NCT01321619
Title: Study Clinical, Multicenter,Phase III,Prospective,Randomized,Comparative Double Blind/Double-dummy to Assess the Efficacy and Tolerability of the Use of Varicell in Reducing the Symptoms Caused by Chronic Venous Insufficiency and Hemorrhoidal Syndrome When Compared With Daflon
Brief Title: Efficacy and Tolerability of the Use of Varicell Compared With Daflon
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vidfarma Indústria de Medicamentos Ltda. (Industry)
Responsible Party: Vidfarma Indústria de Medicamentos Ltda., Industry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VID-VAR-01/11
Record Dates: First submitted 2011-03-15; First posted 2011-03-23 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Venous Insufficiency; Hemorrhoids
Keywords: Chronic venous insufficiency; Hemorrhoidal syndrome; Varicell
MeSH Terms: conditions — Hemorrhoids | interventions — Diosmin; Keratins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varicell (Experimental): Drug A(Varicell) : Administered one tablet three times a day,(oral), the main meals (breakfast, lunch and dinner)for 30 days.
  Interventions: Drug: Daflon
- Placebo daflon (Drug D) (Experimental): Drug D (Placebo Daflon): Administered one tablet two times daily (oral), the main meals (breakfast and dinner)for 30 days.
  Interventions: Drug: Varicell placebo

INTERVENTIONS:
Drug: Daflon — Drug B (Daflon): Administered one tablet two times daily (oral), the main meals (breakfast and dinner)for 30 days.
  Other Names: Diosmin
  Arms: Varicell
Drug: Varicell placebo — Drug C (Varicell placebo) : Administered one tablet three times a day,(oral), the main meals (breakfast, lunch and dinner)for 30 days.
  Other Names: keratin; Circanetten.
  Arms: Placebo daflon (Drug D)

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of Varicell compared to Daflon, in reducing the symptoms caused by chronic venous insufficiency and hemorrhoidal syndrome.

DETAILED DESCRIPTION:
To evaluate the efficacy of Varicell compared with Daflon in the symptomatic treatment of chronic venous insufficiency and hemorrhoidal syndrome.

To evaluate the tolerability of the use of Varicell compared with Daflon in the symptomatic treatment of chronic venous insufficiency and hemorrhoidal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* For both groups
* Patients who consent to participate in the study by signing the Instrument of Consent.
* Patients of all ethnic groups, of both sexes and aged at least 18 years old and maximum 65 years old;
* Being for seven days without any medication or treatment related to the venous system.
* Patients able to make proper use of medication;

For Group V - Chronic Venous Insufficiency.

* Presence of at least two symptoms (pain, heaviness and discomfort) in the lower limbs with scores greater than 3 measured by visual analogue scale;
* Clinical diagnosis of varicose veins rating of 0 to 3 by CEAP;

In Group H - hemorrhoidal syndrome.

* Presence of at least two symptoms (pain in the anorectal evacuation to walk and / or at rest, feeling of anal discomfort (burning, itching, irritation) to evacuate to walk and / or at rest, bloating in the anorectal region, the presence and intensity of bleeding in the anorectal region, the presence and intensity of mucus in the anorectal region) with a score equal to or greater than 3 measured by visual analogue scale;
* Clinical Diagnosis of Hemorrhoids grade 1 and grade 2.

Exclusion Criteria:

Pregnant or lactating;

* Patients aged less than 18 years old or older than 65 years old;
* Patients with a history of hypersensitivity to any component of the formula;
* Use of medications phlebotonics in the last 7 days;
* previous venous surgery;
* Patients with renal and liver failure.
* Patients with gastritis or gastric ulcer;
* Patients with acute inflammatory diseases of the bowel, intestinal obstruction, appendicitis;
* Patients with ileus, stenosis, atony, undiagnosed abdominal symptoms, colonopathy inflammatory abdominal pain of unknown cause dehydration and loss of water and electrolytes and constipation;
* Patients with blood coagulation disorders;
* Any condition which in the opinion of the physician investigator is significant and can make the patient unsuitable for study or that might put you under additional risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Study to evaluate the efficacy and tolerability of the Use of Varicell Compared with Daflon. | 30 days
  Evaluate the efficacy of varicell compared with Daflon in the symptomatic treatment of chronic venous insufficiency and / or hemorrhoidal syndrome.

SECONDARY OUTCOMES:
Study to evaluate the efficacy and tolerability of the Use of Varicell Compared with Daflon. | 30 days
  Evaluate the tolerability of the use of Varicell when used for symptomatic treatment of chronic venous insufficiency and / or hemorrhoidal syndrome compared with Daflon.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Waisberg, Investigator, Principal Investigator — ABC School of Medicine; Walter Campos Júnior, Investigator, Principal Investigator — Edmundo Vasconcelos Hospital Teacher; Laércio Robles, Investigator, Principal Investigator — Santa Marcelina Hospital
Locations (1):
- Santa Marcelina Hospital, São Paulo, São Paulo, Brazil